CLINICAL TRIAL: NCT00824031
Title: Study of Mental Care in Spain
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Esteban Medina. Epidemiology Specialist, AstraZeneca Pharmaceutical
Other Study IDs: NIS-NES-DUM-2008/4
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Schizophrenia
Keywords: schizophrenia; medical mental care; caregiver; Sapin
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Non-interventional, multicenter, cross-sectional study to evaluate the mental care received by schizophrenic patients and their caregivers in Spain irrespective of the drug prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia (DSM-IV criteria)
* Attended to the mental care units for the first time in 2006

Exclusion Criteria:

* Participation in another clinical trial
* Other criteria that according to the medical criteria make difficult the normal development of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged 18-year old or older who has been diagnosed as schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2009-01; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Camberwell's scale of Needs Analysis (CAN) | Once
Caregiver Needs Questionnaire(CNF) | Once

SECONDARY OUTCOMES:
Health of the Nation Outcome Scales (HoNOS) | Once

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Gomez-Beneyto, Study Chair — University of Valencia; Alberto Gonzalez, Study Chair — Hospital Universitario Principe de Asturias
Locations (9):
- Spain (9):
  - Research Site, Ferrol, A Coruna
  - Research Site, Jerez de la Frontera, Cadiz
  - Research Site, Torrejón de Ardoz, Castellon
  - Research Site, Avilés, Principality of Asturias
  - Research Site, La Plana, Valencia
  - Research Site, Bilbao, Vizcaya
  - Research Site, Córdoba
  - Research Site, Girona
  - Research Site, Madrid